CLINICAL TRIAL: NCT06682377
Title: Evaluation of Clinical Efficacy of Radiofrequency Ablation Using Combined RF Energy Delivery Mode and Octopus Electrodes for Hepatocellular Carcinoma: a Prospective Multicenter Study
Brief Title: Radiofrequency Ablation Using Combined RF Energy Delivery Mode and Octopus Electrodes for Hepatocellular Carcinoma
Acronym: SM-OCT-01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-068-1163
Record Dates: First submitted 2024-11-02; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- No touch RFA with dual switching monopolar + bipolar mode (Experimental)
  Interventions: Procedure: Radiofrequency ablation alone

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — No touch RFA with dual switching monopolar + bipolar mode

SUMMARY:
The purpose of this study is to evaluate, through a prospective multicenter trial, the procedural time, safety, technical success rate for achieving a safety margin of at least 5 mm around the tumor, and the clinical efficacy (local and remote recurrence rates: estimated local recurrence rate at 12 months) of radiofrequency ablation using the "No-touch" technique. This approach employs Octopus electrodes and combined radiofrequency energy delivery (dual switching monopolar and bipolar mode) for the treatment of hepatocellular carcinoma.

ELIGIBILITY:
**Inclusion Criteria**

1. Agreement to the protocol requirements and provision of informed consent.
2. Age between 20 and 85 years.
3. Child-Pugh Class A or B7.
4. Patients with liver cirrhosis who are candidates for radiofrequency ablation (RFA) based on multi-detector computed tomography (MDCT) or multi-detector computed tomography (MRI) within 60 days, with a suspected hepatocellular carcinoma (HCC) lesion of 1-3 cm.

   * **HCC Diagnostic Criteria:** A. Presence of risk factors (e.g., hepatitis B virus (HBV) positive, hepatitis C virus (HCV) positive, liver cirrhosis).

   B. Findings consistent with HCC on at least one imaging modality (MDCT, dynamic MRI, or Primovist MRI) according to the Korean Liver Cancer Association (KLCA) criteria.

   C. Histological diagnosis of HCC.
5. No prior history of HCC treatment, or if previously treated, no recurrence confirmed for at least two years.

**Exclusion Criteria**

1. Presence of three or more malignant liver tumors.
2. Diffuse infiltrative type tumors with unclear boundaries.
3. Recurrent HCC within two years of previous treatment.
4. Tumors adhered to major hepatic vessels or bile ducts by more than 5 mm.
5. Poor tumor visibility even with contrast-enhanced ultrasound (CEUS)-fusion image guidance.
6. Vascular invasion by malignant liver tumors.
7. Severe coagulopathy (platelets <50,000/mm³ or International Normalized Ratio (INR) >50% prolongation).
8. Presence of extrahepatic metastasis.
9. Situations where obtaining appropriate data for the study is unlikely.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Estimated local tumor progression rate | 12 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No